CLINICAL TRIAL: NCT00316433
Title: Phase II Study of Oxaliplatin and CPT-11 as First Line Treatment for Extensive Stage Small Cell Lung Cancer
Brief Title: Oxaliplatin/CPT-11 for Extensive Stage Small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Swedish Medical Center (Other)
Collaborators: Sanofi-Synthelabo (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OX-03-099
Record Dates: First submitted 2006-04-18; First posted 2006-04-20 (Estimated); Last update posted 2007-04-05 (Estimated); Status verified 2007-04

CONDITIONS: Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Irinotecan; Oxaliplatin

INTERVENTIONS:
Drug: Irinotecan (CPT-11)
Drug: Oxaliplatin (Eloxatin)

SUMMARY:
The purpose of this study is to determine the safety and effectiveness of the combination of oxaliplatin and irinotecan (CPT-11) in patients with previously untreated, advanced small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated extensive small cell lung cancer
* No prior chemotherapy
* No prior radiotherapy except for the treatment of brain metastases

Exclusion Criteria:

* Prior treatment for extensive stage small cell lung cancer
* Known hypersensitivity to any of the components of oxaliplatin or CPT-11
* Greater than grade 2 peripheral neuropathy
* Known HIV or Hepatitis B or C (active, previously treated or both)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24
Dates: Start 2005-02; Study Completion 2007-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard (Jack) West, MD, Principal Investigator — Swedish Medical Center Cancer Institute
Locations (1):
- Swedish Medical Center Cancer Institute, Seattle, Washington, United States